CLINICAL TRIAL: NCT05357820
Title: A Phase I, Single-center, Open-label, Fixed-sequence Study of AB-106 in Chinese Healthy Adult Men Evaluated the Effects of Itraconazole and Rifampicin on AB-106 Pharmacokinetics
Brief Title: A Study of AB-106 in Chinese Healthy Adult Men Evaluated the Effects of Itraconazole and Rifampicin on AB-106 PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nuvation Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB-106-C110
Record Dates: First submitted 2021-07-09; First posted 2022-05-03 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2022-04

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Itraconazole cohort (Experimental)
  Interventions: Drug: AB-106, Itraconazole
- Rifampicin cohort (Experimental)
  Interventions: Drug: AB-106, Rifampicin

INTERVENTIONS:
Drug: AB-106, Itraconazole — single dose AB-106 at Day1, Itraconazole QD at Day14~Day28, single dose AB-106 at Day17
  Arms: Itraconazole cohort
Drug: AB-106, Rifampicin — single dose AB-106 at Day1, Itraconazole QD at Day14~Day32, single dose AB-106 at Day21
  Arms: Rifampicin cohort

SUMMARY:
AB-106-C110 is China-only study, for investigating the drug interaction between AB-106 and CYP3A4 inhibitor (Itraconazole)/CYP3A4 inducer (Rifampin)（n=56）

ELIGIBILITY:
Inclusion Criteria:

1. The subject is willing to give written informed consent.
2. The subject is capable to communicate well with investigator and comply with comply with protocol throughout the study.
3. Aged between 18 to 55 at giving written informed consent.
4. Chinese male healthy subjects (No clinical abnormality by medical history query, physical examination, vital signs, 12 lead ECG and clinical laboratory test)
5. Body weight greater than 50.0 kg, and body mass index between 19 and 26 kg/m2, inclusive.
6. For fertile males, agree to use effective contraception methods during the study intervention period and for at least 90 days after the last dose of investigational drug, and agree not to donate sperm during this period.

Exclusion Criteria:

1. Any presence or history of clinically significant hematology, nephrology, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, mental, neurological, or allergic diseases (including drug allergy, but not including untreated, asymptomatic seasonal allergies when administered).
2. Any clinically significant laboratory abnormality (hematology, biochemistry [fasting], coagulation, thyroid function, urinalysis.)
3. systolic blood pressure (SBP) < 90 mmHg or ≥140 mmHg, diastolic blood pressure (DBP) < 50 mmHg or ≥ 90 mmHg, and clinically significant abnormality based on the judgment of investigators
4. Any presence or history of eye disease in whom the risk is increased by the participation to the study or treatment with investigational drug in the opinion of the investigator, such as glaucoma, retinal detachment, vitreous turbidity, and moths.
5. The 12-lead ECG showed QTcF > 450 milliseconds (msec) or QRS interval > 120 msec. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times, and the average of 3 QTcF or QRS values should be used to determine subject's eligibility.
6. Fever within 5 days before the administration.
7. Active hepatitis B virus (HBV) surface antigen, hepatitis C virus antibody (HCV Ab), human immunodeficiency virus (HIV) or treponema pallidum (TP) antibody
8. Within 28 days prior to the first dose of study treatment, use of food or drugs that are known potent CYP3A4 inhibitors including (but not limited to) atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, aceto-eandomycin, voriconazole, grapefruit, grapefruit juice, grapefruit, citrus fruits or grapes Pomelo mixed species; or potent CYP3A4 inducers including (but not limited to) carbamazepine, phenobarbital, phenytoin, rifabutin, and rifampin and St. John's wort; or CYP3A4 substrates with narrow therapeutic window including (but not limited to)dihydroergotamine, ergotamine, pimozide, astemizole, cisapride, and terfenadine.
9. Chinese herbal medicine or tonic must be withdrawn at least 28 days prior to the first dose of study treatment; Any clinical study drug is prohibited within 3 months or 5 half-lives prior to the first dose of investigational drug; Any prescription/over-the-counter drug/dietary supplement is prohibited within 14 days or 5 half-lives prior to the first dose of investigational drug; as an exception, acetaminophen/paracetamol can be used at a dose of 1 g/day.
10. Vaccinated with live or attenuated vaccine within 28 days prior to the first dose of study treatment
11. Subject is unwilling to withdraw foods containing caffeine or purines (such as coffee, tea, cola, chocolate) from 48h before first dose to finishing the last PK sample collection.
12. Alcohol intake is greater than 14 units/week (1 unit of alcohol is equivalent to 360 mL of beer, or 150 mL of wine, or 45 mL of baijiu), or subject is unwilling to withdraw alcohol from 48h before first dose to finishing the last PK sample collection.
13. Smoking more than 5 cigarette per day, or subject is unwilling to withdraw nicotine from 48h before first dose to finishing the last PK sample collection.
14. Any drug abuse, or taking any soft drug (such as marijuana) or hard drugs (heroin, cocaine, etc.) from 1 year before and during the study period.
15. Any significant surgical history within 6 months prior to the first dose of study treatment.
16. Blood donation or blood loss ≥ 400 mL within 3 months or ≥ 200 mL within 1 month prior to the first dose of study treatment.
17. Presence of gastrointestinal, liver, kidney disease or other diseases or sequelae that are known to interfere with drug absorption, distribution, metabolism, or excretion. With a history of sensitivity to heparin or heparin-induced thrombocytopenia
18. Unwilling or incapable to follow the lifestyle standard described in the protocol.
19. Staff members of any institution affiliated with the clinical site and their immediate family members. Immediate family members refer to persons with blood or legal relationship, including spouses, children, parents, and siblings.
20. Ineligible to participate in the study based on the judgement of investigators

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
AB-106 PK Exposure Parameters | 29 days
  Peak Plasma Concentration (Cmax)
AB-106 PK Exposure Parameters | 29 days
  Area under the plasma concentration versus time curve (AUC)

SECONDARY OUTCOMES:
AB-106 PK Parameters | 29 days
  Time to drug peak plasma concentration (Tmax)
AB-106 PK Parameters | 29 days
  Percentage of area under the curve from time of the last quantifiable concentration to infinity to area under the curve to infinity (AUC_extr%)
AB-106 PK Parameters | 29 days
  Lambda_z, first-order rate constant associated with the terminal portion of the curve (λz)
AB-106 PK Parameters | 29 days
  Terminal phase elimination half life (t1/2)
AB-106 PK Parameters | 29 days
  Apparent total clearance (CL/F)
AB-106 PK Parameters | 29 days
  Apparent volume of distribution (Vz/F)
Safety Assessment | 47 days
  Adverse events (AEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital of Capital Medical University, Beijing, China